CLINICAL TRIAL: NCT03505294
Title: The Effect of Task-Oriented Training on the Physical and Cognitive Functions in Patients With Multiple Sclerosis
Brief Title: The Effect of Task-Oriented Training in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 229
Record Dates: First submitted 2018-04-19; First posted 2018-04-23 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; task-oriented training; physical performance; cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind trial
Who Masked: Outcomes Assessor
Masking Description: To ensure blinding, the assessor physiotherapist will not be aware of the arm to which the subjects belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-oriented training (Experimental): "Task-oriented training" consisting of 10 different motor tasks will be applied.
  Interventions: Other: Task-oriented training
- Control group (No Intervention): The control group will be taught relaxation exercises and will be asked to perform.

INTERVENTIONS:
Other: Task-oriented training — "Task-oriented training" consisting of 10 different motor tasks including lower extremity and upper extremity activities will be applied to the training group twice a week for 6 weeks.
  Arms: Task-oriented training

SUMMARY:
It is reported that 85% of MS patients have gait disturbance, 87.9% balance, 35-90% fatigue and 45-60% cognitive problems. Rehabilitation approaches based on the motor control systems model, the plasticity concept, the motor learning principles, have been found to be effective for solving these problems. With these rehabilitation approaches, it is aimed to develop the ability of the person to meet the task and environmental demands and to realize the highest quality and the right function with maximum potential by consuming the least energy in different environmental conditions of different tasks. "Task-oriented training" may be one of the most effective among the evidence-based rehabilitation approaches for these goals.

The purpose of this study is to determine the effect of "Task-Oriented Training" on the physical and cognitive functions in patients with multiple sclerosis.

DETAILED DESCRIPTION:
The study was designed as a randomized, controlled, single-blind trial. The patients will be randomly assigned to two groups, the "task-oriented training" group, and the control group. "Task-oriented training" consisting of 10 different motor tasks including lower extremity and upper extremity activities will be applied to the training group twice a week for 6 weeks. The control group will be taught relaxation exercises and will be asked to perform the exercises 2 times for 6 weeks at home.

Statistical analyses will be performed using the SPSS software version 15 (SPSS Inc. Chicago, IL, USA). The pre-training and post-training measurements of groups will be compared with the Wilcoxon Test. The significance level was set at p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are ambulatory and volunteer to participate to the study, in a stable phase of the disease, without relapses in the last 3 month, with an EDSS between 2-5,5.

Exclusion Criteria:

* Participants who have orthopedic, vision, hearing, or perception problems
* Patients who have any cardiovascular or pulmonary disease in which exercise is contraindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Gait Assessment | ten minutes
  The Functional Gait Assessment is a 10-item walking-based balance test, with each item scored 0 to 3. The high score shows that the balance is better.
Walking ability | Five minutes
  The 12-item Multiple Sclerosis Walking Scale (MSWS-12) is a self-assessment scale. During the last 2 weeks 12 problems that can occur during walking due to MS are evaluated (1:no limitation, 5:extreme limitation).
mobility | ten minutes
  Timed Up and Go Test
Modified Sensory Organization Test | Fifteen minutes
  The Modified Sensory Organization Test, which is performed using computerized posturography, measures postural sway in response to 4 different sensory conditions is measured using a force platform.
upper extremity function | ten minutes
  9-Hole Peg Test
cognitive function | thirty minutes
  The Brief Repeatable Battery of Neuropsychological Tests consists of the Selective Reminding Test, the 10/36 Spatial Recall Test, the Symbol Digit Modalities Test, the Paced Auditory Serial Addition Test and the Word List Generation Test.

SECONDARY OUTCOMES:
Balance Scale | ten minutes
  Berg Balance Scale (BBS) rates performance from 0 (cannot perform) to 4 (normal performance) on 14 items. It has shown to be a valid measure with high inter and interrater reliability for people with MS.
Balance Confidence | Five minutes
  Activities-specific Balance Confidence (ABC) is a scale in which the patient rates his perceived level of confidence while performing 16 daily living activities.
Fatigue Severity | five minutes
  In the Fatigue Severity Scale (FSS), participants are asked to rate their fatigue level between 1 and 7 in the 9 statements (including motivation, exercise, physical functioning, carrying out duties, and interfering with work, family, or social life) during the last week.
Fatigue Impact | Five minutes
  Fatigue impact scale consists of forty questions and evaluates the effects of fatigue on the 3 dimensions of daily life activities; cognitive function, physical function and psychosocial function. Each question is graded between 0 (no problem) and 4 (maximum problem).
Physical Activity | ten minutes
  International Physical Activity Questionnaire- Long version (IPAQ) measures total physical activity domains including work-related, transport-related activity, leisure-time, domestic and gardening (yard) activities over the last 7 days. The total scores for each activity type including walking, moderate-intensity activities, and vigorous-intensity activities were calculated by using the answers given to these domains.
Neuropsychological Questionnaire | one minute
  Multiple Sclerosis Neuropsychological Questionnaire (MSNQ) is a self-administered 15-item questionnaire that measure of neuropsychological functioning in everyday life.

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chisari C, Venturi M, Bertolucci F, Fanciullacci C, Rossi B. Benefits of an intensive task-oriented circuit training in Multiple Sclerosis patients with mild disability. NeuroRehabilitation. 2014;35(3):509-18. doi: 10.3233/NRE-141144. PMID 25248447
- [Background] Straudi S, Martinuzzi C, Pavarelli C, Sabbagh Charabati A, Benedetti MG, Foti C, Bonato M, Zancato E, Basaglia N. A task-oriented circuit training in multiple sclerosis: a feasibility study. BMC Neurol. 2014 Jun 7;14:124. doi: 10.1186/1471-2377-14-124. PMID 24906545
- [Background] Salci Y, Fil A, Armutlu K, Yildiz FG, Kurne A, Aksoy S, Nurlu G, Karabudak R. Effects of different exercise modalities on ataxia in multiple sclerosis patients: a randomized controlled study. Disabil Rehabil. 2017 Dec;39(26):2626-2632. doi: 10.1080/09638288.2016.1236411. Epub 2016 Oct 29. PMID 27794631
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Walker ML, Austin AG, Banke GM, Foxx SR, Gaetano L, Gardner LA, McElhiney J, Morris K, Penn L. Reference group data for the functional gait assessment. Phys Ther. 2007 Nov;87(11):1468-77. doi: 10.2522/ptj.20060344. Epub 2007 Sep 4. PMID 17785375
- [Background] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Background] Oxford Grice K, Vogel KA, Le V, Mitchell A, Muniz S, Vollmer MA. Adult norms for a commercially available Nine Hole Peg Test for finger dexterity. Am J Occup Ther. 2003 Sep-Oct;57(5):570-3. doi: 10.5014/ajot.57.5.570. PMID 14527120
- [Background] Boringa JB, Lazeron RH, Reuling IE, Ader HJ, Pfennings L, Lindeboom J, de Sonneville LM, Kalkers NF, Polman CH. The brief repeatable battery of neuropsychological tests: normative values allow application in multiple sclerosis clinical practice. Mult Scler. 2001 Aug;7(4):263-7. doi: 10.1177/135245850100700409. PMID 11548987
- [Background] Benedict RH, Munschauer F, Linn R, Miller C, Murphy E, Foley F, Jacobs L. Screening for multiple sclerosis cognitive impairment using a self-administered 15-item questionnaire. Mult Scler. 2003 Feb;9(1):95-101. doi: 10.1191/1352458503ms861oa. PMID 12617275
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Armutlu K, Keser I, Korkmaz N, Akbiyik DI, Sumbuloglu V, Guney Z, Karabudak R. Psychometric study of Turkish version of Fatigue Impact Scale in multiple sclerosis patients. J Neurol Sci. 2007 Apr 15;255(1-2):64-8. doi: 10.1016/j.jns.2007.01.073. Epub 2007 Mar 6. PMID 17337007
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694